CLINICAL TRIAL: NCT03849911
Title: EEG and SEP Evaluation for Good and Poor Neurological Prognosis After Cardiac Arrest: a Prospective Multicenter Cohort Trial (proNeCA)
Brief Title: EEG and SEP Evaluation for Good and Poor Neurological Prognosis After Cardiac Arrest
Acronym: ProNeCA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Antonello Grippo, Grippo Antonello, MD, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: AOU Careggi
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Neurological Prognosis Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurophysiological Prognosis — SEP and EEG evaluation for Neurological Prognosis of Cardiac Arrest
Diagnostic Test: Multimodal Prognosis for poor early neurological outcome — Brain CT, SEP and EEG evaluation

SUMMARY:
Hypoxic-Ischemic-encephalopathy (HIE) is a severe and frequent neurological complication of successful cardiopulmonary-resuscitation after cardiac arrest (CA). Prognosticating neurological outcomes in patients with HIE is challenging and recent guidelines suggest a multimodal approach. Only few studies have analyzed the prognostic power of the association between instrumental tests and, in addition, most of them were monocentric, retrospective and evaluating only poor outcome.

DETAILED DESCRIPTION:
Post-anoxic encephalopathy is a severe and frequent neurological complication of successful cardiopulmonary resuscitation and it is usually responsible for coma onset in patients surviving a CA. A reliable early assessment of the neurological prognosis is an important research goal because it could address CA patient management within intensive care units (ICUs).

However, prognosticating neurological outcomes in patients with HIE is challenging and recent guidelines suggest a multimodal approach. Only few studies have analyzed the prognostic power of the association between instrumental tests and, in addition, most of them were monocentric, retrospective and evaluating only poor outcome.

Thus, the investigators designed a multicenter prospective cohort study to assessing the prognostic power of the association of electroencephalogram(EEG) and somatosensory evoked potentials(SEPs) for the prediction of both poor and good neurological outcomes at different times after CA.

The principal aim of this study will be to evaluate the prognostic power of EEG performed in comatose patients within the first 12h after CA for good outcome prediction (cerebral performance categories CPC 1-2-3) and to evaluate its prognostic power for the poor outcome prediction (CPC 4-5) when performed at 24 and 72h after CA.

Moreover, the investigators will aim to evaluate if the combination of EEG and SEPs will allow to correctly identify a greater number of patients with both poor and good outcomes (when performed within the first 12h) and with poor outcomes (when performed after 72h) compared with the use of only a single test. In addition, the investigators will evaluate if the concordance of EEG/SEP patterns will increase the prognostic reliability obtained with a single test.

Finally, the investigators will aim to confirm if the prognostic power of the bilaterally absent(AA) SEP pattern for poor outcome prediction will be reliable at any time of recording after CA, and if other SEP pathological patterns will assume an analogous ominous prognostic significance.

ADDENDUM: after the conclusion of the enrollment we investigated the availability of brain CT data obtained within the first 24 hours after CA. In 7 over 13 centers, including the coordinator center (AOU Careggi, Florence) early brain CT data were available.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 18 and 90 years of age and
* comatose patients surviving after CA with a Glasgow Coma Scale (GCS) <9

Exclusion Criteria:

* patients with surgical or traumatic causes of CA,
* patients showing contemporary presence of other neurological diseases (i.e. traumatic brain injury or brain infarction),
* patients with previous severe neurological diseases,
* patients with remote pathological anamnesis showing severe diseases with life expectancy less than 6 months,
* patients with previous severe disability,
* contemporary presence of confounding factors that hamper clinical evaluation (in particular the consciousness state)
* patients with contemporary absence of cortical response N20/P25 and lemniscal wave P14

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every major patient after CA admitted to the follow intensive care unit: Careggi University Hospital (Firenze), which will be the coordinating center, San Giuseppe Hospital (Empoli), Bufalini Hospital (Cesena), Santa Maria delle Croci Hospital (Ravenna), Santa Maria NuovaHospital (Reggio Emilia), Ospedale Civile of Baggiovara (Baggiovara-Modena),Maggiore Hospital of Lodi (Lodi-Milano),San Raffaele Hospital (Milano), Ospedale Civile of Legnano (Legnano-Milano), Policlinico Umberto Primo (Roma), Santa Maria della Misericordia Hospital (Perugia), San Salvatore Hospital (L'Aquila), Galliera Hospital (Genova)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Cerebral Performance Categories | Month 6
  Neurological outcome will be the primary outcome measure and it will be assessed at 6 months after CA using CPC as follows: CPC 1, no or minor neurological deficits; CPC 2, moderate disability; CPC 3, severe disability; CPC 4, unresponsive wakefulness state and CPC 5, death. Neurological outcome will be dichotomized into 'good' (CPC 1-3) and 'poor' (CPC 4-5) outcomes

SECONDARY OUTCOMES:
Electroencephalography, EEG | hour: 12-24-72
  American Clinical Neurophysiology Society (ACNS) EEG terminology
Somatosensory Evoked Potentials, SEP | hour: 12-24-72
  According to the cortical responses of each hemisphere
Brain CT | within 24 hours
  Caudate nucleus(CN), putamen(PU) and posterior limb of the internal capsule(PIC) were bilaterally identified as circular (0.6cm2) regions of interest(ROIs) where density measurement (Hounsfield Units-HU) were performed. At the corpus callosum(CC) level, the density value was considered the same bilaterally. The GM/WM ratio at basal ganglia level was calculated as follows: GM/WM ratio= (CN+PU)/(CC+PIC)

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scarpino M, Lolli F, Lanzo G, Carrai R, Spalletti M, Valzania F, Lombardi M, Audenino D, Contardi S, Grazia Celani M, Marrelli A, Mecarelli O, Minardi C, Minicucci F, Politini L, Vitelli E, Peris A, Amantini A, Grippo A, Sandroni C; ProNeCA Study Group. Do changes in SSEP amplitude over time predict the outcome of comatose survivors of cardiac arrest? Resuscitation. 2022 Dec;181:133-139. doi: 10.1016/j.resuscitation.2022.10.025. Epub 2022 Nov 12. PMID 36375653